CLINICAL TRIAL: NCT03616301
Title: Open-label, Randomized, Crossover, Two-period, Two-sequence, Single-center, Comparative Bioequivalence Study of Clavamox, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml (Pharmtechnology LLC, Belarus), and Augmentin®, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml (GlaxoSmithKline Trading CJSC, Russia), in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Clavamox, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml (Pharmtechnology LLC, Belarus), and Augmentin®, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml (GlaxoSmithKline Trading CJSC, Russia), in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FRM-04-AMOX version 2.0
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-07

CONDITIONS: Bioequivalence
Keywords: bioequivalence; amoxicillin; clavulanic acid; Augmentin
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is an open-label study; the subjects and the investigator will not be blinded towards the identity of the study products. However, analysts will be blinded towards identity of the study products administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clavamox, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml (Experimental): Clavamox, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml is the test product. 14 of 28 subjects in each of two cohorts (total number of enrolled volunteers - 56) will be given single oral dose (5 ml containing 400 mg of amoxicillin and 57 mg of clavulanic acid) in period 1 and period 2 of the clinical part of the study.
  Interventions: Drug: Clavamox
- Augmentin®, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml (Active Comparator): Augmentin®, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml is the reference product. 14 of 28 subjects in each of two cohorts (total number of enrolled volunteers - 56) will be given single oral dose (5 ml containing 400 mg of amoxicillin and 57 mg of clavulanic acid) in period 1 and period 2 of the clinical part of the study.
  Interventions: Drug: Augmentin®

INTERVENTIONS:
Drug: Clavamox — Clavamox, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml, manufactured by Pharmtechnology LLC, Belarus
  Arms: Clavamox, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml
Drug: Augmentin® — Augmentin®, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml, marketed by CJSC GlaxoSmithKline Trading, Russia
  Arms: Augmentin®, Powder for Oral Suspension, 400 mg + 57 mg / 5 ml

SUMMARY:
This is an open-label, randomized, single-center, single-dose, two-treatment, two-sequence, two-period, crossover, comparative study, where each subject will be randomly assigned to the reference or the test formulation in each period of the study (sequences RT or TR), in order to evaluate if both formulations are bioequivalent.

DETAILED DESCRIPTION:
The objective of this study is to establish if two formulations of amoxicillin + clavulanic acid combination are bioequivalent. Also monitoring, registration and evaluation of adverse events will be performed. The test formulation is Clavamox, powder for oral suspension, 400 mg + 57 mg / 5 ml (Pharmtechnology LLC, Belarus). The reference formulation is Augmentin®, powder for oral suspension, 400 mg + 57 mg / 5 ml (GlaxoSmithKline Trading CJSC, Russia).

56 healthy adult volunteers of both genders, with age ranging from 18 to 45 years old, will be divided into two cohorts with equal number of subjects (28). Each subject in a cohort will receive single dose (5 ml containing 400 mg of amoxicillin and 57 mg of clavulanic acid) of the test or the reference formulation with 200 ml of water after an overnight fast of at least 10 hours, according to the pre-defined randomization list, i. e. 14 subjects in each cohort will receive the test product and 14 subjects in each cohort will receive the reference product. Subjects will fast 4 hours after administration of the study drugs during each study period. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour prior to administration of the study drugs and 2 hours after administration of the study drugs in each period.

In each period blood samples will be collected before dosing and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing (total number: 19). The washout period is 7 days.

A validated HPLC/MS/MS method will be used to determine plasma concentrations of two analytes (amoxicillin and clavulanic acid).

ANOVA will be performed on log-transformed pharmacokinetic parameters Cmax, AUC0-t and 90% confidence interval will be constructed for the ratio of geometric least square means of the test and the reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval for each analyte, both falls within the acceptable range of 80.00% to 125.00% for Cmax and AUC0-t.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men or women aged between 18 to 45 years
* subjects having no clinically significant medical history and no clinically significant abnormalities in general physical examination, laboratory assessments and imaging studies.
* body mass index 18.5-29.9 kg/m² with body mass >45 kg and ≤100 kg
* non-breastfeeding women
* non-pregnant women
* if subject is a female and is of child bearing potential, she should be practicing an acceptable non-hormonal method of birth control for the duration of the study(at least 14 days before the start of the study, throughout the study and 14 days after the completion of the study), such as a combination of male condom and diaphragm with spermicide
* if subject is a male and and has a female partner of child bearing potential, he should be practicing an acceptable method of birth control for the duration of the study(at least 14 days before the start of the study, throughout the study and 14 days after the completion of the study), such as a combination of male condom and spermicide (double barrier method).
* subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations.

Exclusion Criteria:

* Subjects with a known history of allergic disorders.
* Hypersensitivity to the active substances, to any of the penicillins or to any of the excipients of the test and the reference product.
* Subjects with a known history of drug intolerance.
* History of a severe immediate hypersensitivity reaction (e.g. anaphylaxis) to any of beta-lactam agents (e.g. a cephalosporin, carbapenem or monobactam).
* History of jaundice/hepatic impairment due to amoxicillin/clavulanic acid.
* Dehydration due to diarrhea, vomiting or other reasons within 24 hours prior to start of the first period of the study.
* Subjects with history of psychiatric disorders.
* History of convulsions, epilepsy and any other neurological disorders.
* Dietary sodium restriction within two weeks prior to start of the study or adherence to special types of diets (vegetarian, vegan, with salt restriction) and lifestyle (work at night, extreme physical activity).
* Use of gestagen-containing injectable hormonal contraceptives, implants, intrauterine hormonal therapeutic systems within 6 months prior to start of the study.
* Female subjects of child bearing potential having unprotected intercourse with an unsterilized sexual partner within 30 days prior to start of the study.
* Consumption of xanthine-containing foods and drinks (tea, coffee, coca-cola, chocolate) within 72 hours prior to start of the first period of the study.
* Consumption of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including cranberry juice and other cranberry drinks) within 14 days prior to start of the study.
* Cardiovascular, respiratory, gastrointestinal diseases, neuroendocrine disorders, renal and/or hepatic impairment, blood system disorders.
* Other conditions which, according to the researcher's judgment, may affect absorption, distribution, biotransformation and elimination of any formulation or increase risks of deterioration of volunteer's condition.
* Surgical interventions on the gastrointestinal tract with the exception of appendectomy.
* Acute infectious diseases less than 4 weeks prior to the start of the study.
* ECG abnormalities.
* Sitting systolic blood pressure < 100 mm Hg or > 130 mm Hg and/or sitting diastolic blood pressure < 70 mm Hg or > 90 mm Hg.
* Heart rate <60 or >80 beats per minute at screening check-in.
* Use of liver enzyme inducers and inhibitors, in particular isoenzyme CYP3A4 (inducers: omeprazole, cimetidine, products containing the extract of Hypericum perforatum, barbiturates, carbamazepine, phenytoin, glucocorticoids; inhibitors: antiviral drugs, clarithromycin, ciprofloxacin, gestodene) within 30 days prior to the start of the study.
* Use of any systemic drugs within 14 days prior to the start of the study.
* Use of OTC drugs, including herbs and nutritional supplements within 7 days prior to the Dosing Date. (including vitamins and natural food additives, phyto supplements,herbal preparations such as, cat's claw, angelica officinalis, oenothera, feverfew, garlic, ginger, ginkgo, red clover, horse chestnut, green tea, ginseng).
* Donation of plasma or blood (450 ml or more) within 2 months prior to the start of the study.
* Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine or 50 ml of spirits) or history alcoholism, drug addiction, drug abuse.
* Smoking more than 10 cigarettes per day.
* Participation in other clinical trials of medicines within 3 months prior to the start of the study.
* Positive test for syphilis, hepatitis B, hepatitis C or HIV.
* Positive pregnancy test (for female subjects with child bearing potential).
* Breast-feeding.
* Positive test for alcohol.
* Positive urinary screen test for drugs of abuse.
* Oral contraceptives should be withdrawn 2 months prior to the start of the study.
* Subjects who refuse to comply with the study protocol and/or not credible therein and who are, at the discretion of the Principal Investigator, unable to understand and assess the information about the study, expected risks and possible discomfort in the process of signing written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Cmax of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to the last measured concentration
Cmax of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to the last measured concentration

SECONDARY OUTCOMES:
Number of treatment-related adverse events (AE) for the test and the reference products as assessed by guidance predefined in the protocol | 17 days
  An AE is defined as any untoward medical occurrence in a subject administered an investigational product and which does not necessarily have a causal relationship with the treatment. The data from participants who had taken at least one investigational product was analyzed.
AUC0-∞ of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to to infinite time
AUC0-∞ of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to to infinite time
Tmax of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Time to maximum measured plasma concentration
Tmax of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Time to maximum measured plasma concentration
T1/2 of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Elimination or terminal half-life
T1/2 of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Elimination or terminal half-life
Kel of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Elimination rate constant
Kel of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Elimination rate constant
AUCresid of amoxicillin for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Residual area
AUCresid of clavulanic acid for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0.25, 0.5, 0.75, 1.00, 1.25, 1.5, 1.75, 2.00, 2.33, 2.67, 3.00, 3.5, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00 hours after dosing
  Residual area

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Professor, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- State Autonomous Healthcare Facility of the Yaroslavl Region "Clinical Hospital No. 2", Yaroslavl, Yaroslavl Oblast, Russia